CLINICAL TRIAL: NCT06904456
Title: Advanced HIV Disease During the First Six Months on Antiretroviral Therapy in Zambia
Acronym: AHD-Zambia
Status: Recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Clinton Health Access Initiative Inc. (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: H-45653; INV-031690 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2025-03-23; First posted 2025-04-01 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Advanced HIV Disease
Keywords: Antiretroviral therapy (ART); Zambia; Service delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1. Prospective cohort: Cohort 1 is a prospective cohort of adults screened for AHD during the approximately three-month data collection period of the AHD Zambia study. Clients will be enrolled into the study if they 1) are not on ART or have been on ART for up to one month, and 2) are screened for AHD on the day of study enrollment or, if missed on the day they are screened for AHD, will be enrolled at the next clinic visit within one month of AHD screening. Record review for up to 12 months before and 12 months after study enrollment. Baseline survey and qualitative follow up.
- 2. Hybrid cohort: Cohort 2 is a hybrid cohort of all adult HIV clients recorded in study sites' AHD screening registers, improvised registers, and/or clinic records as having been screened for AHD at or before ART initiation in the 12 months preceding the start of Cohort 1 data collection. Electronic and paper medical record data will be collected for all of Cohort 2 for the 12 months before and 12 months after the AHD screening date. A subset of Cohort 2 respondents-those who return to the study sites for a clinic visit during the data collection period-will be invited to consent and participate in a quantitative survey and in follow-up qualitative interviews, similar to Cohort 1 enrollees.
- 3. Inpatient cohort: Cohort 3 includes adult HIV clients admitted in a study health facility for AHD management. Under the Zambia Ministry of Health's "hub and spoke model" for AHD management, AHD patients requiring hospitalization are admitted to hub facilities. Of the 24 study facilities in AHD-Zambia, 8 are hubs that admit AHD patients. The remaining 16 study sites refer AHD clients requiring admission to the nearest hospital. We will enroll Cohort 3 only at the 8 sites that offer inpatient admission for AHD.
- 4. Provider cohort: At each study site, we will ask the facility manager to refer us to up to 5 staff who provide care for AHD clients and represent different cadres. This may include doctors and clinical officers, nurses, counselors, and pharmacists, though we anticipate the majority of respondents to be doctors, nurses and clinical officers, who provide most HIV care in Zambia. Each cohort participant will be administered a one-time survey regarding AHD care at the facility.

SUMMARY:
In Zambia, an estimated 20% of HIV-positive clients continue to present for first-time antiretroviral therapy (ART) initiation or re-initiation with advanced HIV disease (AHD). The Zambia Ministry of Health (MOH) and other key stakeholders lack information about the characteristics and behaviors of AHD clients, including how they are defined and diagnosed (e.g. low CD4 count v. clinical condition), their demographic and socioeconomic profiles, their HIV care histories, what services they receive, and their short-term outcomes (achieve viral suppression, remain AHD, disengage from care, die) and the timing of these outcomes.

The Retain6 project aims to improve HIV treatment outcomes during clients' first six months on ART, when disengagement from care and mortality are highest. This protocol, called Advanced HIV disease during the first six months on antiretroviral therapy in Zambia (AHD Zambia), describes an observational study that will describe the experiences of clients who are diagnosed with AHD upon ART initiation (or re-initiation) in Zambia. Data collected will include clinical and socioeconomic characteristics, clinical and non-clinical needs, services delivered and received, and clients' and providers' concerns and preferences. The study's overall goal is to provide information to the Zambia MOH, treatment program partners, providers, and other stakeholders to better understand who is presenting with AHD in Zambia, how they are currently managed, and their treatment outcomes after starting ART. This information will be useful in determining interventions and guideline changes that might improve short- and long-term outcomes for AHD patients.

The study, which will be conducted in collaboration with the Zambia MOH, will include retrospective file reviews, prospective quantitative surveys with outpatient and inpatient clients, qualitative focus group discussions (FGDs) and interviews with clients, and provider surveys and interviews.

ELIGIBILITY:
Cohort 1

Inclusion

* ≥18 years old
* Presenting at a study site clinic for HIV diagnosis or care
* Not currently on ART (or on ART for up to 1 month if enrolled at next visit after AHD screening)
* Screened for AHD by clinic, prior to or within 1 month of ART initiation
* Written informed consent to participate

Exclusion

* Pregnant and/or presenting for antenatal care
* Too ill at the time of AHD screening and at the next clinic visit to participate in the study
* Unable to communicate in any of the languages into which the questionnaire has been translated or that is known to the research assistant

Cohort 2

Inclusion

* ≥18 years old
* Living with HIV and screened for AHD at a study site within 12 months of the start of study prospective data collection at that site
* All inclusion criteria for the full cohort
* Initiated/re-initiated ART within the past 6 months
* Returns to the study site for a clinic visit during the study enrollment period
* Written informed consent to participate

Exclusion

* Pregnant and/or presenting for antenatal care as reported in records
* All exclusion criteria for the full cohort
* Too ill at the time of study enrollment visit to participate in the study
* Unable to communicate in any of the languages into which the questionnaire has been translated or that is known to the research assistant
* Been on ART >6 months

Cohort 3

Inclusion

* ≥18 years old
* Living with HIV
* Admitted for inpatient care related to AHD
* Initiated or re-initiated ART within the last 6 months
* Written informed consent to participate

Exclusion

* Pregnant and/or presenting for antenatal care
* Not physically, mentally, or emotionally able to participate in the study prior to discharge, in the opinion of facility or study staff
* Unable to communicate in any of the languages into which the questionnaire has been translated or that is known to the research assistant
* Confined to tuberculosis isolation ward; intensive care unit; or other ward specifically for clients with acute infectious disease.

Cohort 4

Inclusion

* Employed by or at the study site for at least 6 months
* Directly interact with clients presenting with AHD
* Written informed consent to participate

Exclusion

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be adult HIV treatment patients and providers at the study sites who meet inclusion and exclusion criteria for each cohort.
Sampling Method: Non-Probability Sample
Enrollment: 11800 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Initiation characteristics | 6 months
  Characteristics of clients presenting with AHD at treatment initiation or re-initiation, compared to clients screened but found not to have AHD.
Inpatient characteristics | 6 months
  Characteristics of clients admitted to hospital after an AHD diagnosis.
Six-month retention | 6 months
  Retention in care of clients presenting with AHD at 6 months after AHD diagnosis.
Six-month viral suppression | 6 months
  Viral suppression of clients presenting with AHD at 6 months after AHD diagnosis.

SECONDARY OUTCOMES:
12-month retention | 12 months
  Retention in care of clients presenting with AHD at 12 months after AHD diagnosis.
12-month viral suppression | 12 months
  Viral suppression of clients presenting with AHD at 12 months after AHD diagnosis.
Guideline fidelity | 12 months
  Facility and provider fidelity to Zambia's AHD guidelines
Costs | 12 months
  Costs of resources used to provide AHD care

CONTACTS AND LOCATIONS:
Overall Officials: Thandiwe Ngoma, Principal Investigator — CHAI-Zambia
Locations (1):
- CHAI-Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymized data generated by the study, such as survey responses and qualitative data (not routine medical record data, which will not be owned by the study team), will be posted to a public data repository after final closure of the study protocol.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available after study protocol closure. Data will remain in the public repository in perpetuity.
Access Criteria: Data will be public (fully dis-identified) using the public data repository.

REFERENCES:
- [Derived] Ngoma T, Kamanga A, Scott N, Morgan A, Reddy Marri A, Makwalu T, Mulenga L, Sivile S, Benade M, Haimbe P, Shakwelele H, Rosen S. Advanced HIV disease during the first six months on antiretroviral therapy in Zambia: research protocol for a prospective, observational, multi-cohort study. Gates Open Res. 2025 Aug 27;9:66. doi: 10.12688/gatesopenres.16359.1. eCollection 2025. PMID 40896557
- See also: repository for study publications and reports — https://sites.bu.edu/ambit/retain6-resources/